CLINICAL TRIAL: NCT00480584
Title: A Phase I Trial of GemCap-T, Capecitabine in Combination With Gemcitabine and Erlotinib (Tarceva®) in Patients With Advanced Pancreatic Adenocarcinoma
Brief Title: A Phase I Trial of Capecitabine in Combination With Gemcitabine and Erlotinib for Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14624; OSI3482s (Other: Genentech)
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Metastatic Pancreatic Carcinoma
Keywords: pancreatic; gemcitabine; erlotinib (HER1/epidermal growth factor receptor [EGFR] tyrosine kinase inhibitor); capecitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Capecitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GemCap-T Dose Escalation (Experimental): GemCap-T, capecitabine in combination with gemcitabine. Dose Escalation 6 Cycles @ 28 Days.
  Interventions: Drug: gemcitabine; Drug: capecitabine; Drug: erlotinib

INTERVENTIONS:
Drug: gemcitabine — Levels 1 through 4: 1000 mg/m^2
  Other Names: Gemzar®
Drug: capecitabine — Level 1: 500 mg/m^2; Level 2: 825 mg/m^2; Level 3: 1000 mg/m^2; Level 4: 1250 mg/m^2
  Other Names: Xeloda
Drug: erlotinib — Levels 1 through 4: 100 mg
  Other Names: Tarceva®

SUMMARY:
This is a phase I clinical trial examining the safety, feasibility, and toxicity of gemcitabine and erlotinib when given in combination with capecitabine in adult patients with locally advanced unresectable or metastatic pancreatic adenocarcinoma.

Treatment will be administered at Moffitt on an outpatient basis and consists gemcitabine once per week for 3 weeks, followed by a week off treatment. Erlotinib (tablet) taken by mouth continuously starting with day one of cycle 1 with capecitabine taken twice per day on days 1-14 of each cycle followed by a 2 week off treatment rest period. An accelerated dose-escalation scheme will be employed with 4 planned dose levels. Whenever patients have been enrolled at a given dose with at most 1 DLT, the protocol will be stopped and the dose will be called the maximum tolerated dose (MTD). Patients will be treated at the recommended phase II dose (RPTD) to confirm tolerability at that dose.

In the absence of treatment delays due to adverse events, treatment may continue for 6 cycles or until disease progression and patients may continue on the study regimen unless they experience an adverse event that meets the criteria for a dose limiting toxicity.

DETAILED DESCRIPTION:
This is a phase I clinical trial examining the safety, feasibility, and toxicity of gemcitabine and erlotinib when given in combination with capecitabine in adult patients with locally advanced unresectable or metastatic pancreatic adenocarcinoma. This combination of drugs has never been used before.

Screening tests will consists of demographics, a medical history, and physical exam, vital signs, height, weight, performance status, blood counts, chemistries, and clotting. There will also be an electrocardiogram (EKG), tumor measurement (computed tomography [CT Scan] or magnetic resonance imaging [MRI] or positron emission tomography CT [PET-CT]), cancer antigen (CA 19-9), and a serum pregnancy test (for women of childbearing potential). Tumor measurements are also performed after cycle 2, 4, and 6 (study end).

Treatment will be administered on an outpatient basis and consists of both intravenous (IV) medication and tablets taken by mouth. The gemcitabine will be administered at Moffitt once per week for 3 weeks, followed by a week off treatment. One tablet of erlotinib will be taken by mouth continuously starting with day one of cycle 1 while capecitabine will be taken twice per day on days 1-14 of each cycle followed by a 2 week off treatment rest period. This set of treatments is called a cycle. One full cycle of treatment will last 28 days and a total of 6 cycles of treatments are planned. Before each cycle we will repeat the blood counts and a brief physical exam (vital signs) will be recorded weekly during the first 3 weeks of the 28 day cycle of treatment (when receiving Gemcitabine).

An accelerated dose-escalation scheme will be employed with 4 planned dose levels. Patients will be enrolled at the lowest dosage level, if no patients have unacceptable toxicity, the dose will be escalated and additional patients enrolled. If one of the patients at a given dose level experiences a dose limiting toxicity (DLT), more patients will be treated at that dose level. When 2 patients have DLTs at the same dose, the dose will be deescalated to the previous dose and additional patients will be enrolled. After de-escalation begins, whenever patients have been enrolled at a given dose with at most 1 DLT, the protocol will be stopped and the dose will be called the maximum tolerated dose (MTD). Patients will be treated at the recommended phase II dose (RPTD) to confirm tolerability at that dose.

In the absence of treatment delays due to adverse events, treatment may continue for 6 cycles or until disease progression. Patients may continue on the study regimen unless they experience an adverse event that meets the criteria for a dose limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic adenocarcinoma that is metastatic or unresectable.
* Previously untreated with chemotherapy in the metastatic setting. Prior 5-fluorouracil (5-FU) or capecitabine treatment is allowed if: 1) it was given as part of a combined modality chemoradiation regimen and 2) no greater than 30% of bone marrow was included in the field and 3) the treatment free interval has been > 6 weeks
* Must have measurable disease, defined as at least one lesion that can be measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* Age greater than or equal to 18 years
* Because no dosing or adverse event data are currently available on the use of capecitabine in combination with gemcitabine and erlotinib in patients <18 years of age, children are excluded from this study. Pancreatic adenocarcinoma is primarily a disease of the elderly.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) less than or equal to 2 (Karnofsky greater than or equal to 60%).
* Life expectancy > 8 weeks
* Must have normal organ and marrow function as defined below:

  1. leukocytes, greater than or equal to 3,000/μl
  2. absolute neutrophil count, greater than or equal to 1,500/μl
  3. platelets, greater than or equal to100,000/μl
  4. total bilirubin, less than or equal to 2.5 X institutional upper limit of normal
  5. AST(SGOT)/ALT(SGPT), less than or equal to 2.5 X institutional upper limit of normal (ULN)
  6. AST(SGOT)/ALT(SGPT), less than or equal to 5 X institutional ULN in patients with liver metastasis
  7. creatinine, less than or equal to 1.5 X institutional ULN
  8. creatinine clearance, > 30 ml/min (Cockcroft-Gault method)
* Has a negative serum or urine pregnancy test within 7 days prior to initiation of therapy (female patients of childbearing potential).
* Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Patients will agree to continue contraception for 30 days from the date of the last study drug administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior chemotherapy for pancreatic adenocarcinoma in the metastatic setting are not eligible.
* Chemoradiation within the last 6 weeks prior to registration are not eligible
* Known allergy or severe reactions to gemcitabine, capecitabine, or tyrosine kinase inhibitors are not eligible
* May not be receiving any other investigational agents or received investigational agents within the 28 days prior to registration.
* Known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events.
* Prior malignancy in the last 3 years, except basal cell carcinoma, squamous cell, or in-situ cervical cancer
* ECOG PS 3-4
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because gemcitabine and capecitabine are Class D agents with the potential for teratogenic or abortifacient effects.
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, human immunodeficiency virus (HIV) positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with erlotinib or other agents administered during the study.
* Creatinine clearance < 30 ml/min (Cockcroft-Gault method)
* Patients that require ongoing (chronic) treatment with medications metabolized by CYP3A4 (saquinavir, ritonavir, nelfinavir, indinavir, ketoconazole, itraconazole, nefazodone, clarithromycin, atazanavir, rifampicin, rifabutin, rifapentine, phenytoin, carbamazepine, phenobarbital, St. John's Wort) who cannot be switched to alternate medications that are not metabolized by CYP3A4 are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Within 4 months of Cycle 1 Day 1 (C1D1)
  The Maximum-tolerated dose (of capecitabine) is determined as the dose level at which two or more of six patients experience dose-limiting toxicity. The MTD will not exceed 1250 mg/m2.

SECONDARY OUTCOMES:
Recommended Phase II Dose (RPTD) | Within 4 months of Cycle 1 Day 1 (C1D1)
  To determine the recommended phase II dose (RPTD)of capecitabine when given in combination with gemcitabine and erlotinib. The recommended phase 2 dose is determined as the highest dose level below the MTD where 0-1 out of 6 patients have dose limiting toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Springett, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States